CLINICAL TRIAL: NCT01377766
Title: Study of Psychological Factors on the Occurence of Bell's Palsy
Brief Title: The Relationship Between Psychological Factors and Bell's Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); Xiangyang No.1 People's Hospital (Other); Renmin Hospital of Wuhan University (Other); Fudan University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Yichang Hospital of Traditional Chinese Medicine (Other); The First Hospital of Hebei Medical University (Other); Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Wei Wang, Department of Neurology and Psychology, Tongji Hospital, Huazhong University of Science and Technology
Other Study IDs: 2006CB504502-3
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Bell's Palsy
Keywords: Bell's palsy; psychological stress; personality factors; psychological factors
MeSH Terms: conditions — Bell Palsy; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study was to explore the risk factors for Bell's palsy (BP) and to examine whether psychological factors are the potential risk factors for the occurrence of BP.

DETAILED DESCRIPTION:
We conducted a case-control, multi-center clinical investigation. A total of 695 subjects were assigned to the case group (n=355) and the control group (n=340). All the BP patients were enrolled from 11 State Hospitals in China, and all the controls were selected from the same district to match for the patients. The study was coordinated by a tertiary referral centre, Tongji Hospital. The House-Brackmann grading system and Facial Disability Index (FDI) was adopted to assess the BP patients. Kessler 10-Item Psychological Distress Scale（K10）was usde to explore the psychological distress, and the Cattell 16 Personality Factor (16PF) scale was employed to evaluate the personality profiles of all subjects.

ELIGIBILITY:
Inclusion criteria:

1. Patients who were diagnosed to have unilateral facial-nerve weakness without any identifiable causes within 168 hours after onset of symptoms;
2. aged 18 to 65 years.

Exclusion criteria：

1. illiterate;
2. the facial paralysis is caused by herpes zoster;
3. recurrent facial paralysis;
4. noticeable asymmetry of the face before the illness which may affect the evaluation;
5. history of peptic ulcer disease, severe hypertension, uncontrolled diabetes, liver and kidney dysfunction, pregnancy, mental illness, or serious systemic diseases which may affect the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 695 subjects were assigned to Cases Group (n=355) and Control Group (n=340).
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann scale (HBS) | within 168 hours after onset of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Institute of Integrated Traditional Chinese and Western Medicine, Wuhan, Hubei, China